CLINICAL TRIAL: NCT00702208
Title: The Feasibility and Acceptability of Using the Delphi Screener for Cervical Cytology Testing Among Low Income Women in New York City
Brief Title: Feasibility of Delphi Screener for Cervical Cytology
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Delphi Devices BV (Unknown)
Responsible Party: Principal Investigator, Carolyn L. Westhoff, Professor of Obstetrics and Gynecology, Population and Family Health and Epidemiology at the New York-Presbyterian Hospital at the Columbia University Medical Center, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AAAD1382
Record Dates: First submitted 2008-05-30; First posted 2008-06-20 (Estimated); Results first posted 2014-01-13 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2013-07

CONDITIONS: Cervical Neoplasia
Keywords: cervical cytology; Pap smear; self-sampling; abnormal; normal
MeSH Terms: conditions — Antisocial Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm study (Other): Paired laboratory results for clinician-collected and Screener collected specimens for cytology (and high-risk human papillomavirus testing for sub-sample)
  Interventions: Device: Delphi Screener

INTERVENTIONS:
Device: Delphi Screener — Self-sampling device for cervical vaginal lavage
  Other Names: Pantarhei Screener; Mermaid

SUMMARY:
The aim of this study is to see whether a new self-sampling device, the Delphi Screener (Delphi Devices, Scherpenzeel, Netherlands), can be used for cervical cancer screening. The results using the new device will be compared to results using the current gold standard. The gold standard is clinician-collected endo-cervical and ecto-cervical specimens (often referred to as a 'Pap smear'). Additionally, women will be asked about the acceptability of using the device and how easy it is to understand the user instructions.

The Delphi Screener is a sterile, plastic, syringe-like device containing buffered saline which allows a woman to collect her own vaginal lavage (to 'self-squirt'). The hypothesis is that the device may work well for cervical cytology and will be acceptable to the women in the study.

ELIGIBILITY:
Inclusion Criteria:

* Valid Pap smear in last 1-3 months obtained at participating clinic
* 18 years or older
* Self-report being able to read in English and/or Spanish
* Willing to sign informed consent

Exclusion Criteria:

* Used vaginal product (douche, spermicide, antifungal) in last 48 hours
* Last menses started ≤ 4 days prior to enrollment visit
* No uterus / history of hysterectomy
* Self-report currently pregnant
* Self-report currently breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Westhoff, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Presbyterian Hospital, New York, New York, United States

REFERENCES:
- [Derived] Jones HE, Mansukhani MM, Tong GX, Westhoff CL. Validity and reliability of using a self-lavaging device for cytology and HPV testing for cervical cancer screening: findings from a pilot study. PLoS One. 2013 Dec 20;8(12):e82115. doi: 10.1371/journal.pone.0082115. eCollection 2013. PMID 24376516

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from cervical cancer screening patients from three ambulatory clinics at the New York Presbyterian Hospital from December 1, 2008 to August 31, 2009.
Pre-assignment Details: Eligiblity criteria for participation were: 18 years of age or older, not currently pregnant, not currently breastfeeding, self-reported comfort reading in English or Spanish or their own. Women were scheduled to attend the clinic to use the self-lavaging device 1-3 months after their standard-of-care cervical cancer screening.
Groups:
- Single Arm Study of Delphi Screener: Paired laboratory results for clinician-collected and Screener collected specimens for cytology (and high-risk HPV testing for sub-sample)
  All women were asked to self-collect a cervicovaginal lavage using the Screener during the enrollment study visit. The entire visit took approximately 30-40 minutes. Women generally took 5-10 minutes to self-lavage on their own in a private room.
Period: Overall Study
Arm/Group | Single Arm Study of Delphi Screener
Started | 198
Completed | 167
Not Completed | 31
Not completed — Lost to Follow-up | 28
Not completed — Did not self-lavage | 1
Not completed — Unsatisfactory colposcopy | 2

BASELINE CHARACTERISTICS:
Groups:
- Single Arm Study: Paired laboratory results for clinician-collected and Screener collected specimens for cytology (and high-risk HPV testing for sub-sample)
Arm/Group | Single Arm Study
Number analyzed (Participants) | 198
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 195
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 198

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity
Description: We calculated sensitivity of self-collected lavage with cytology to detect histologically confirmed high grade lesions (cervical intraepithelial neoplasia, CIN, 2+); specificity for histology-negative (CIN 1 or lower), paired cytology negative, or a third cytology negative; and kappa for paired results.
  The cytology specimens were collected 1-3 months apart and women with abnormal results for cytology were followed through January 2010 for final histology endpoints.
Time Frame: 1-3 months between 2 specimen collections
Measure: Number (95% Confidence Interval); unit: % of participants correctly diagnosed
Groups:
- Single Arm Study of Delphi Screener: Paired laboratory results for clinician-collected and Screener collected specimens for cytology (and high-risk HPV testing for sub-sample)
Arm/Group | Single Arm Study of Delphi Screener
Number analyzed (Participants) | 167
% of participants correctly diagnosed
  sensitivity | 0.86 [0.42 to 1.00]
  specificity | 0.80 [0.73 to 0.96]

2. Secondary Outcome: Outcome: Acceptability of Device
Description: On a visual analog scale from 0-10 cm, preference for clinician-collected specimen (0) vs. self-lavage specimen (10) for future cervical cancer screening
Time Frame: cross-sectional - asked at time of Screener use
Population: For acceptability, 197 women used the device; 30 of these women did not have valid gold standard results but did respond to acceptability, thus for acceptability endpoint the sample size is 197 (while the sample size is 167 for sensitivity, specificity and kappa analyses due to insufficient sepcimens /loss to follow-up for colposcopy).
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Single Arm Study of Delphi Screener
Number analyzed (Participants) | 197
units on a scale | 9.6 [7.1 to 9.9]

3. Primary Outcome: Kappa Coefficient
Description: Kappa comparing clinician-collected cytology result to self-lavage cytology result
Time Frame: 1-3 months between 2 specimen collections
Measure: Number (95% Confidence Interval); unit: kappa coefficient for paired specimens
Arm/Group | Single Arm Study of Delphi Screener
Number analyzed (Participants) | 167
kappa coefficient for paired specimens | 0.36 [0.25 to 0.47]

ADVERSE EVENTS:
Arm/Group | Single Arm Study
Serious Adverse Events (participants affected / at risk) | 0/198
Other Adverse Events (participants affected / at risk) | 0/198

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No